CLINICAL TRIAL: NCT03993262
Title: A Multicenter Randomized, Controlled, Double-blinded Trial to Evaluate Efficacy and Safety of Bortezomib in Patients With Severe Autoimmune Encephalitis
Brief Title: Trial to Evaluate Efficacy and Safety of Bortezomib in Patients With Severe Autoimmune Encephalitis
Acronym: Generate-Boost
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jena University Hospital (Other)
Collaborators: Federal Ministry of Education and Reserach (BMBF) (Unknown)
Responsible Party: Principal Investigator, Christian Geis, Prof. Dr. med., Jena University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZKSJ0120; 2024-514494-21-00 (EU CTIS Number); 2019-001423-12 (EudraCT Number); DRKS00017497 (Registry Identifier: DRKS); 01GM1908E (Registry Identifier: Funding code BMBF (Federal Ministry for Education and Research))
Record Dates: First submitted 2019-06-12; First posted 2019-06-20 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Autoimmune Encephalitis
Keywords: autoimmune disease; autoimmune encephalitis; bortezomib; NMDAR; LGI1; encephalitis
MeSH Terms: conditions — Autoimmune Diseases of the Nervous System; Autoimmune Diseases; Encephalitis | interventions — Bortezomib

STUDY DESIGN:
Intervention Model Description: 1:1 randomization will be done centrally and stratified by site. Block randomization of variable block sizes will be used.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study drug will be provided blinded by the local pharmacy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Interventional (Experimental): 1 to 3 cycles Bortezomib with 1,3mg/m2 body surface s.c. + 20mg dexamethasone p.o. on days 1, 4, 8 and 11 (= 1 cycle)
  Interventions: Drug: Bortezomib
- Placebo (Placebo Comparator): 1 to 3 cycles placebo (NaCl solution) s.c. + 20mg dexamethasone p.o. on days 1, 4, 8 and 11 (= 1 cycle)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bortezomib — 1 to 3 cycles Bortezomib with 1,3mg/m2 body surface s.c. + 20mg dexamethasone p.o. on days 1, 4, 8 and 11 (= 1 cycle)
  Arms: Interventional
Drug: Placebo — 1 to 3 cycles placebo (NaCl solution) s.c. + 20mg dexamethasone p.o. on days 1, 4, 8 and 11 (= 1 cycle)
  Other Names: isotonic NaCl solution
  Arms: Placebo

SUMMARY:
Autoimmune Encephalitis is a disorder of the central nervous system caused by bodily substances, called antibodies. Antibodies normally help the body to prevent infections. However, in this disorder, the antibodies turn against the body itself and especially against cells in the brain and disturb the normal brain function. They are therefore called autoantibodies.

There is no specific therapy for patients with autoimmune encephalitis so far. At the moment, the symptoms are treated with approved medications such as cortisone and immunotherapies also used in oncology. These therapies are unspecified and aim to reduce the number of autoantibodies and to contain the autoimmune process. In this trial we aim to test a new therapy option: in this therapy the body cells producing autoantibodies will be specifically targeted by a substance called bortezomib.

The trial addresses patients with severe autoimmune encephalitis. The aim of the trial is to evaluate the efficacy and safety of bortezomib in patients with severe autoimmune encephalitis.

DETAILED DESCRIPTION:
Autoimmune encephalitis is characterized by autoantibodies against neuronal surface antigens like the NMDA (N-methyl-D-aspartate) receptor or LGI1 (Leucin-rich glioma inactivated protein 1). So far, no specific therapy exists for this disease. Actual treatment includes combination therapies aiming for a reduction of pathogenic antibodies and containing the autoimmune process. In first line, patients are treated with plasmapheresis and cortisone. In second line, Rituximab and/or cyclophosphamide are administered. The response to these treatments are, however, often delayed and insufficient.

Therefore, we need a specific therapy aiming at the antibody-producing plasma cells.

Bortezomib is a proteasome inhibitor which interferes with NF-kB (nuclear factor kB) and the ubiquitin proteasome signaling pathway. Bortezomib acts preferably on cells with high protein synthesis - like plasma cells - and induces cell death in these cells. Bortezomib is used since more than a decade in chemotherapy of the multiple myeloma. Additionally, it is reported for systemic autoimmune diseases like lupus erythematodes that bortezomib leads to a depletion of plasma cells and therefore reduces the number of pathogenic antibodies and improves clinical outcome. The therapeutic potential of bortezomib for NMDAR encephalitis is described in a first case series with 5 patients.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed severe autoimmune encephalitis (defined as mRS ≥ 3) with autoantibodies to neuronal surface proteins in cerebrospinal fluid and / or serum
* Pretreatment with rituximab
* Age ≥18 years
* signed informed consent
* Women of childbearing potential (up to 2 years after menopause): negative pregnancy test

Exclusion Criteria:

* pregnancy/breast-feeding
* acute infiltrative pulmonary and pericardial disease
* malignant tumor under current chemotherapy
* Simultaneous participation in another intervention study
* Previous participation in this study
* Known hypersensitivity to an ingredient of the investigational product
* Continued therapy with glucocorticoids / rituximab during the study duration (last dose must be administered before the first dose of the investigational product)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-05-13 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
modified Rankin-Score (mRS) | 17 weeks after first administration of the study drug
  modified Rankin-Score from 0 = no symptoms to 6 = death

SECONDARY OUTCOMES:
modified Rankin-Score (mRS) | 3, 6, 9 and 13 weeks after first administration of the study drug; GCS Score also 17 weeks after first administration of the study drug
  modified Rankin-Score from 0 = no symptoms to 6 = death
Length of in-hospital stay / length of ICU stay | until 17 weeks after first administration of the study drug
  Number of days in hospital or on ICU for each patient from first administration of the study drug until 17 weeks after first administration of the study drug
Immune response | at study start and 17 weeks after first administration of the study drug
  Antibody titer (in serum and liquor) and cellular immune response (FACS analysis of liquor)
neurocognitive function assessed by Montreal Cognitive Assessment | at study start and 17 weeks after first administration of the study medication
  total score of the Montreal Cognitive Assessment (MoCA) (0 to max. 30 points = best possible result)
neurocognitive function assessed by Mini-Mental Status Test | at study start and 17 weeks after first administration of the study medication
  total score of the Mini-Mental Status Test (MMST) (0 to max 30 points = best possible result)
neurocognitive function assessed by Rey Auditory Verbal Learning Test | at study start and 17 weeks after first administration of the study medication
  total score of the Rey Auditory Verbal Learning Test (RAVLT) (memory performance assessed by 3 word lists which are read to the patient and should be recalled and repeated by the patient; different proceeding for the 3 word lists)
neurocognitive function assessed by Neuropsychiatric Inventory Questionnaire | at study start and 17 weeks after first administration of the study medication
  total score of the Neuropsychiatric Inventory Questionnaire (NPI) (0 = best score to max 36 (patient) or 60 (caregiver)
safety of Bortezomib regarding polyneuropathy, increase of liver enzymes and secondary infections | until 17 weeks after first administration of the study drug
  number of polyneuropathy cases, number of increased liver enzymes, number of secondary infections
safety of Bortezomib regarding polyneuropathy | until 17 weeks after first administration of the study drug
  number of polyneuropathy cases
safety of Bortezomib regarding increase of liver enzymes | until 17 weeks after first administration of the study drug
  number of increased liver enzyme values
Secondary infections due to Bortezomib | until 17 weeks after first administration of the study drug
  number of secondary infections
Hematotoxicity events due to Bortezomib | until 17 weeks after first administration of the study drug
  number of hematotoxicity events
Gastrointestinal toxicity due to Bortezomib | until 17 weeks after first administration of the study drug
  number of gastrointestinal toxicity events
total Glasgow Coma Scale (GCS) | 3, 6, 9, 13 and 17 weeks after first administration of the study drug
  GCS from 3 to 15 points (sum of 3 subscores eye response (1 to 4 points), motor response (1 to 6 points), verbal response (1 to 5 points); highest score = best score; 1= worst score)
Destruction marker UCH-L1 (Ubiquitin carboxy-terminal hydrolase L1) in serum and liquor | at baseline visit and 17 weeks after first administration of the study drug
  Analysis of destruction marker UCH-L1 in serum and liquor
Destruction marker Neurofilament light chain (in serum and liquor) | at baseline visit and 17 weeks after first administration of the study drug
  Analysis of destruction marker Neurofilament light chain in serum and liquor
Destruction markers GFAP (glial fibrillary acidic protein) in serum and liquor | at baseline visit and 17 weeks after first administration of the study drug
  Analysis of destruction marker GFAP in serum and liquor
Destruction marker TAU proteins in serum and liquor | at baseline visit and 17 weeks after first administration of the study drug
  Analysis of destruction marker TAU in serum and liquor

CONTACTS AND LOCATIONS:
Overall Officials: Christian Geis, Prof., Study Director — University Hospital Jena
Locations (17):
- Germany (17):
  - Ludwig-Maximilians-Universität München, Klinikum Großhadern, München, Bavaria
  - Universitätsklinikum Würzburg, Würzburg, Bavaria
  - Universitätsklinikum Jena, Sektion Translationale Neuroimmunologie, Klinik für Neurologie, Jena, Germany
  - Medizinische Hochschule Hannover, Hanover, Niedersachen
  - Charité - Universitätsmedizin Berlin, Klinik für Neurologie mit Experimenteller Neurologie, Berlin
  - Ruhr-Universität Bochum, St. Josef Hospital, Klinik für Neurologie, Bochum
  - University Hospital Düsseldorf, Clinic for Neurology, Düsseldorf
  - Universitätsklinikum Erlangen, Neurologische Klinik, Erlangen
  - Universitätsklinikum Essen (AöR), Klinik für Neurologie, Essen
  - University Hospital Frankfurt (Main), Clinic for Neurology, Frankfurt
  - Universitätsmedizin Göttingen Georg-August-Universität, Klinik für Neurologie, Göttingen
  - Universitätsmedizin Greifswald, Klinik und Poliklinik für Neurologie, Greifswald
  - Klinik für Neurologie UKSH, Campus Kiel, Kiel
  - Universitätsklinikum Leipzig, Klinik und Poliklinik für Neurologie, Leipzig
  - Universitätsmedizin Mainz, Klinik und Poliklinik für Neurologie, Mainz
  - Universitätsklinikum Münster Klinik für Neurologie, Münster
  - Universitätsklinikum Ulm, Klinik für Neurologie Neurologische Ambulanz, Ulm

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet decided in which way and which data exactly will be shared with other researchers.

REFERENCES:
- [Derived] Wickel J, Chung HY, Platzer S, Lehmann T, Pruss H, Leypoldt F, Gunther A, Scherag A, Geis C; GENERATE Study Group. Generate-Boost: study protocol for a prospective, multicenter, randomized controlled, double-blinded phase II trial to evaluate efficacy and safety of bortezomib in patients with severe autoimmune encephalitis. Trials. 2020 Jul 8;21(1):625. doi: 10.1186/s13063-020-04516-7. PMID 32641101